CLINICAL TRIAL: NCT06178263
Title: Adherence to an Exercise and Healthy Diet Program in Patients With Coronary
Brief Title: Adherence to an Exercise and Healthy Diet Program in Patients With Coronary Heart Disease Aged ≥ 60 Years
Acronym: RE-Start60+
Status: Completed | Type: Observational
Sponsor: University Medicine Greifswald (Other)
Collaborators: German Center of Cardiovascular Diseases (DZHK) (Unknown)
Responsible Party: Sponsor
Other Study IDs: BB138/17
Record Dates: First submitted 2023-11-30; First posted 2023-12-20 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Coronary Heart Disease; Risk Reduction Behavior; Adherence, Treatment
Keywords: physical activity; nutrition; views on ageing; adherence; intervention
MeSH Terms: conditions — Coronary Disease; Risk Reduction Behavior; Treatment Adherence and Compliance; Motor Activity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of the study is to implement a multimodal lifestyle intervention over 3 months in individuals ≥ 60 years of age with coronary heart disease and to examine the adherence to this intervention program. The intervention focus on three main themes: physical activity, healthy nutrition and, if necessary, smoking. The framework is formed by a psychological component: views on ageing.

DETAILED DESCRIPTION:
Long-term adherence to a healthy lifestyle that promotes heart health (e.g. physical activity, healthy diet, non-smoking) is not yet sufficiently achieved in patients with coronary artery disease (≥ 60 years).

Individuals in this study will participate in a 3-month multimodal intervention program. The program includes group and individual sessions with a focus on exercise training and healthy nutrition. Positive views on ageing have been shown to be associated with a healthier lifestyle. Therefore, it seems important to consider views on ageing as part of a lifestyle intervention.

The intervention program starts with a group session containing information on (i) views on ageing and its association to lifestyle and (ii) how to cope with the diagnosis of coronary heart disease in everyday life.The physical exercise training and nutrition intervention will be carried out at least twice a week for at least 60 minutes each and for a period of 3 months. During this time, participants will receive instructions to exercise regularly and adjust their nutrition according to the recommendations. The physical exercise training and nutritional recommendations should be implemented at home. Study participants who smoke tobacco will be motivated to participate in a smoking cessation program. If they are not willing to do this, short, motivating interviews on smoking cessation will be offered.

A pilot study will be conducted using a pre-post design. Patients will be followed over time and data will be collected on anthropometrics, blood samples, cardiopulmonary exercise tests, and 7-day accelerometry at baseline and at 3- and 12-month follow-ups.

ELIGIBILITY:
Inclusion Criteria:

* age of ≥ 60 years
* established CVD defined by a stenosis of ≥ 70% of a least one coronary vessel
* optimal treatment according to the European Society of Cardiology guidelines (2016)

Exclusion Criteria:

* heart failure, left ventricular ejection fraction (LVEF) < 40%
* implanted cardioverter/defibrillator or pacemaker
* recent cardiovascular event ≤ 2 months prior to study inclusion (acute myocardial infarction, resuscitation, re-vascularization, device implantation, or stroke)
* planned coronary revascularization
* uncontrolled blood pressure (systolic blood pressure of ≥ 200 mmHg)
* body mass index ≥ 35 kg/m2
* baseline cardiopulmonary exercise test results precluding safe exercise training (e.g., ischemia or arrhythmias)
* no ability to participate in exercise training (e.g., COPD GOLD III-IV, claudication ≥ 2b, or previous disabling stroke)
* current mental disorder requiring inpatient treatment
* current addictions (excluding tobacco use), florid psychoses, current severe depressive episode (according to ICD-10)
* severe cognitive or physical impairment
* no serious co-existing diseases (e.g., cancer) with life expectancy < 1 year
* weekly self-reported PA ≥ 150 minutes on a moderate intensity level ≤ 6 months prior to study inclusion

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Inpatients at the cardiology ward at Greifswald University Medical Center are asked to take part in the lifestyle intervention study. Eligible patients aged ≥ 60 years will be invited to participate in the study by mail. In order to be included as a study participant, written informed consent is required.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Adherence to a multi-behavioral intervention program | Over 12 weeks (Baseline - 3-months)
  Investigation on (long-term) adherence to a 3-months multi-behavioral intervention program (exploratory); Measures: Documentation list of adherence to supervised physical exercise training program sessions, educational nutrition sessions, and views of ageing sessions.
Feasibility of a multi-behavioral intervention program | Over 12 weeks (Baseline - 3-months)
  Investigation on the feasibility of the 3-months multi-behavioral intervention program (exploratory); Measures: Views of participants about study quality process (semi-structured interview guide including self-developed items; qualitative and quantitative)

SECONDARY OUTCOMES:
Cardiopulmonary exercise testing | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in a parameter of cardiopulmonary exercise testing (VO²max); Measures: standardized measurement of cardiopulmonary exercise testing according to a modified Jones protocol; VO²max in ml O²/min/kg
Obesity marker | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in an abdominal obesity marker (waist circumference); Measures: standardized measurements of waist circumference in cm
Physical behavior by self-report | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in physical behavior; Measures: assessement via questionnaire (Swiss Physical Activity Questionnaire, SWISSPAQ; DOI: https://doi.org/10.4414/smw.2013.13752); questionnaire includes 19 activities and 2 open answers for activities not listed. Patients had to specify the frequency (in times per week), duration (in minutes) and intensity (Borg's subjective rating of perceived exertion) of the activities that they performed in a typical week in the previous 2 months. Metric: MET-hours.
Physical behavior by accelerometry (if valid data are available) | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in physical behavior; Measures: objective measurement of physical behavior by 7-day accelerometry
Smoking by self-report | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in smoking; Measures: assessement via two self-reported items
Cardiometabolic marker (I) | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in plasma triglycerides (in mmol/l); Measures: standardized blood sampling
Cardiometabolic marker (II) | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in high-density lipoprotein cholesterol (in mmol/l); Measures: standardized blood sampling
Cardiometabolic marker (III) | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in glucose (in mmol/l); Measures: standardized blood sampling
Brain-derived neurotrophic factor (BDNF) | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in BDNF (in ng/ml); Measures: standardized blood sampling
Blood pressure | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in blood pressure; Measures: standardized measurements of mean blood pressure (in mmHg)
Views on ageing | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in views on ageing; Measures: assessement via questionnaire (Individual views on ageing: specific (physical loss, social loss, personal growth, gains) and global)
Cardiac anxiety | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in cardiac anxiety; Measures: assessement via questionnaire (Cardiac Anxiety Questionnaire, CAQ; DOI: 10.1016/s0005-7967(99)00132-1); 18-item, three subscales (Fear, 8 items; Avoidance, 5 items; Attention, 5 items). Each item is rated on a 5-point Likert scale with scores ranging from 0 (never) to 4 (always). A high score indicates a greater number of symptoms, greater frequency, or both.
Nutrition | Changes from baseline (vs. 3-months and 12-months follow-up)
  Investigation on changes in nutrition; Measures: assessement via questionnaire (Mediterranean Diet Adherence Screener, MEDAS; doi: 10.1186/s12885-017-3337-y); 14 item, the MEDAS score can range between 0 and 14

CONTACTS AND LOCATIONS:
Overall Officials: Sabina Ulbricht, Prof. Dr., Study Chair — Department of Preventive Research and Social Medicine, University Medicine Greifswald
Locations (1):
- Department of Preventive Resaerch and Social Medicine, Institute for Community Medicine, University Medicine Greifswald, Greifswald, Germany

REFERENCES:
- [Result] Ullrich A, Wenzel K, Bahls M, Voigt L, Konemann S, Dorr M, Wurm S, Ulbricht S. Preliminary results of the cross-sectional associations of sedentary behavior and physical activity with serum brain-derived neurotrophic factor in adults with coronary heart disease. Sci Rep. 2022 Nov 16;12(1):19685. doi: 10.1038/s41598-022-23706-8. PMID 36385629